CLINICAL TRIAL: NCT04452201
Title: Parent Communication for Feeding an Infant With a Heart Defect - Pilot Intervention Study
Brief Title: Parent Communication for Feeding an Infant With a Heart Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-0718; Protocol Version 6/27/2017 (Other: UW Madison); A545000 (Other: UW Madison); NUR/FACULTY (Other: UW Madison)
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Communication; Heart Defects, Congenital; Infant Conditions
Keywords: Communication; Parents; Infants; Congenital Heart Disease; Feeding; Caregiving; Guided Participation
MeSH Terms: conditions — Communication; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Participation (GP) (Experimental): A GP intervention is participatory formal and informal education to support learning of a practice beyond what could occur as efficiently and effectively without guidance. GP uses strategies for teaching-learning that make best use of the family's situation and opportunities, tailored to the parents' needs. The overall goal of the GP intervention is to support parent couples in effectively communicating for parenting work, including care-giving and maintaining the couple's relationship
  Interventions: Behavioral: Guided Participation
- Usual Care (UC) (No Intervention): The UC group will receive standard of care

INTERVENTIONS:
Behavioral: Guided Participation — GP couples' participation together in development of communication competencies in the context of infant care will be supported by a handbook and telephone guidance structured for collaboration with the nurse/research assistant beginning at approximately 2 weeks of age. Two face-to-face sessions are expected prior to hospital discharge, followed by 5 or 6 monthly phone sessions. If the baby is inpatient at the time an intervention session is to take place, the session may be done face-to-face, if more convenient than a phone session for the parents.
  Other Names: GP
  Arms: Guided Participation (GP)

SUMMARY:
The purpose of this study is to pilot test an innovative, guided participation (GP) intervention to help parents develop competencies in communication for parenting an infant with a complex congenital heart defect (CCHD) through the first six months of age.

DETAILED DESCRIPTION:
Study aims are to:

* Investigate the intervention feasibility (capability of being done, carried out, and objectives accomplished), accessibility, acceptability, usefulness, safety, and cost.
* Explore the effect of the GP intervention on outcomes within and between groups and over time.

Sample and Groups:

Parents will be recruited to the study either following a prenatal or postnatal diagnosis of a complex congenital heart defect. 36 families will be recruited and then computer randomized to either the GP or usual care (UC) groups in a 2:1 ratio, with a goal of 30 families completing the study (20 GP families, 10, UC families). Six of the families will be enrolled at American Family Children's Hospital (Madison, WI) (AFCH), with the rest enrolled at CHW. Each participating parent couple will receive an electronic tablet that will be the couple's to keep. A library of published materials from the UW-Health Sciences Library about infant care has been installed on the Tablets for both groups.

GP couples' participation together in development of communication competencies in the context of infant care will be supported by a handbook that is installed on the tablet as well as being given to parents in hard copy, and by telephone guidance, structured for collaboration with the nurse/research assistant beginning at approximately 2 weeks of age. Two face-to-face sessions are expected prior to hospital discharge, followed by 5 or 6 monthly phone sessions. If the baby is inpatient at the time an intervention session is to take place, the session may be done face-to-face, if more convenient than a phone session for the parents.

For both GP and UC groups, data will be collected prior to the infant's discharge from the hospital and at 2 and 6 months after the infant's birth. Two severity of infant illness scores will be computed by a pediatric cardiologist, the first for the neonatal period and the second when the infant is 6 months old. The data collections plus a monthly phone call to learn about infant and family changes make the UC group an attention control group.

A survey regarding use of the materials supplied as part of the study and the couple's communication will be collected at 4 time points from parents in both groups. Baseline and soon after the baby begins oral feeding (up to to one week, both before hospital discharge) and, 2 months and 6 months (both at home, 6 months is end of study).

Each data collection visit will include:

* self-report surveys
* assessment of heart-rate variability (HRV)
* an initial 20-minute interview about what the parents are experiencing and working on as parents, how they are managing stressors, and how caregiving is going
* an infant feeding of usual length
* an approximately 30-minute interview concerning the parents' internal working model of feeding, parenting communication and co-parenting pattern
* a couple problem-solving session with two 7-minute problems, each followed by independent evaluation of the problem session by each parent
* following each visit, data will be obtained from the infant's electronic health record

  * anthropometric data (weight, length, head circumference)
  * illness and treatments
  * medical procedures
  * neurodevelopmental progress

The feeding and the problem solving will be video recorded for in-laboratory coding.

ELIGIBILITY:
Inclusion Criteria:

* Parent couples will be married or partnered (living together),
* English speaking and reading
* Infants will have a CCHD diagnosed by the first week of life, requiring palliative or reparative surgery within the baby's first year

Exclusion Criteria:

* Families will be excluded if either parent is not willing to participate, or is unable to participate due to a communication barrier
* Families will be excluded if either parent is known to have a mental illness that interferes with day-to-day functions or a substance use problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Iowa Family Interaction Rating Scales (IFIRS) scores to measure family dynamics | month 2
  The IFIRS is an Observational macrocoding system where recorded interviews are coded and each code is given a single score upon review. Scores are 1-9 where 1 indicates that the behavior did not occur and 9 indicates the behavior almost always occurs. Families were scored on the following codes at 2 and 6 months: goal setting, problem solving, negotiating issues, and emotion regulating during problem solving.
Iowa Family Interaction Rating Scales (IFIRS) scores to measure family dynamics | month 6
  The IFIRS is an Observational macrocoding system where recorded interviews are coded and each code is given a single score upon review. Scores are 1-9 where 1 indicates that the behavior did not occur and 9 indicates the behavior almost always occurs. Families were scored on the following codes at 2 and 6 months: goal setting, problem solving, negotiating issues, and emotion regulating during problem solving.

SECONDARY OUTCOMES:
Parent-Child Early Relational Assessment (ERA) Scores | up to one week
  The ERA is an observational measure of parental mental attunement and sensitivity and responsiveness to the infant and of the infant's responsive and regulated behavior during feeding. The mean score for each of the six subscale scores are reported: Parental Positive Affective Involvement, sensitivity, & Responsiveness; Parental Negative Affect and behavior (a higher score indicates less of the parental negative affect and behavior); Infant Positive Affect & Communicative and Social Skills; Infant Dysregulation and Irritability; Dyadic Mutuality and Reciprocity; Dyadic Tension. Each item is rated on a 1-5 scale. Five indicates adaptive behavior. Scores may be treated as follows: 4-5 indicates behavior that is positive and of no clinical concern; 3 indicates there is some clinical concern about the behavior; 1-2 indicates behavior of clinical concern.
Parent-Child Early Relational Assessment (ERA) Scores | 2 months
  The ERA is an observational measure of parental mental attunement and sensitivity and responsiveness to the infant and of the infant's responsive and regulated behavior during feeding. The mean score for each of the six subscale scores are reported: Parental Positive Affective Involvement, sensitivity, & Responsiveness; Parental Negative Affect and behavior (a higher score indicates less of the parental negative affect and behavior); Infant Positive Affect & Communicative and Social Skills; Infant Dysregulation and Irritability; Dyadic Mutuality and Reciprocity; Dyadic Tension. Each item is rated on a 1-5 scale. Five indicates adaptive behavior. Scores may be treated as follows: 4-5 indicates behavior that is positive and of no clinical concern; 3 indicates there is some clinical concern about the behavior; 1-2 indicates behavior of clinical concern.
Parent-Child Early Relational Assessment (ERA) Scores | 6 months
  The ERA is an observational measure of parental mental attunement and sensitivity and responsiveness to the infant and of the infant's responsive and regulated behavior during feeding. The mean score for each of the six subscale scores are reported: Parental Positive Affective Involvement, sensitivity, & Responsiveness; Parental Negative Affect and behavior (a higher score indicates less of the parental negative affect and behavior); Infant Positive Affect & Communicative and Social Skills; Infant Dysregulation and Irritability; Dyadic Mutuality and Reciprocity; Dyadic Tension. Each item is rated on a 1-5 scale. Five indicates adaptive behavior. Scores may be treated as follows: 4-5 indicates behavior that is positive and of no clinical concern; 3 indicates there is some clinical concern about the behavior; 1-2 indicates behavior of clinical concern.
Infant Heart Rate Variability | up to 6 weeks
  Infant heart rate variability is a measure of infant physiologic and bio-behavioral regulation.

OTHER OUTCOMES:
Infant Length | up to 6 weeks
Infant Weight | up to 6 weeks
Infant Head Circumference | up to 6 weeks
Bayley III assessment Scores | 6 months
  Each scale (Motor, Cognitive, Language) is assessed and treated separately. The Motor score includes fine and gross motor sub-test scores. The Cognitive score assesses cognitive development. The Language subscales are for assessment of expressive and language development. Scales are scored to a metric with a mean of 100, standard deviation of 14, and range from 40 to 160. A higher score indicates better development. A score below 85 indicates clinical concern.
Satisfaction with Life Scale (SWLS) | baseline
  Quality of life was assessed using the SWLS. The SWLS is a 5-item survey, each item is scored on a 7 point likert scale where 1 is 'strongly disagree' and 7 is 'strongly agree'. The total possible range of scores is 7-35. Higher total scores indicate more satisfaction in life.
Satisfaction with Life Scale (SWLS) | up to one week
  Quality of life was assessed using the SWLS. The SWLS is a 5-item survey, each item is scored on a 7 point likert scale where 1 is 'strongly disagree' and 7 is 'strongly agree'. The total possible range of scores is 7-35. Higher total scores indicate more satisfaction in life.
Satisfaction with Life Scale (SWLS) | 2 months
  Quality of life was assessed using the SWLS. The SWLS is a 5-item survey, each item is scored on a 7 point likert scale where 1 is 'strongly disagree' and 7 is 'strongly agree'. The total possible range of scores is 7-35. Higher total scores indicate more satisfaction in life.
Satisfaction with Life Scale (SWLS) | 6 months
  Quality of life was assessed using the SWLS. The SWLS is a 5-item survey, each item is scored on a 7 point likert scale where 1 is 'strongly disagree' and 7 is 'strongly agree'. The total possible range of scores is 7-35. Higher total scores indicate more satisfaction in life.
Cutrona Social Provisions Scale | baseline
  Parental Relationship Quality was measured using the Cutrona Social Provisions Scale. This is a 24-item self report assessment, each item scored on a 4 point likert scale where 1 is 'strongly disagree' and 4 is 'strongly agree'. The range of total possible scores is 24-96.
Cutrona Social Provisions Scale | up to one week
  Parental Relationship Quality was measured using the Cutrona Social Provisions Scale. This is a 24-item self report assessment, each item scored on a 4 point likert scale where 1 is 'strongly disagree' and 4 is 'strongly agree'. The range of total possible scores is 24-96.
Cutrona Social Provisions Scale | 2 months
  Parental Relationship Quality was measured using the Cutrona Social Provisions Scale. This is a 24-item self report assessment, each item scored on a 4 point likert scale where 1 is 'strongly disagree' and 4 is 'strongly agree'. The range of total possible scores is 24-96.
Cutrona Social Provisions Scale | 6 months
  Parental Relationship Quality was measured using the Cutrona Social Provisions Scale. This is a 24-item self report assessment, each item scored on a 4 point likert scale where 1 is 'strongly disagree' and 4 is 'strongly agree'. The range of total possible scores is 24-96.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Pridham, PhD, RN, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - American Family Children's Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified data collected during the trial, including parents' interview data; coded infant feeding skills; growth and development data; summary measures for heart-rate variability, and parent-child relationship assessment item scores. Researchers, including doctoral students in nursing, whose proposed use of the data for subsequent clinical research has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months after publication of primary outcomes, and ending 5 years after that date.
Access Criteria: Proposals should be directed to kpridham@wisc.edu. If approved after review by regulatory counsel, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.

REFERENCES:
- [Background] Pridham K, Brown R, Clark R, Limbo RK, Schroeder M, Henriques J, Bohne E. Effect of guided participation on feeding competencies of mothers and their premature infants. Res Nurs Health. 2005 Jun;28(3):252-67. doi: 10.1002/nur.20073. PMID 15884024
- [Background] Pridham KF, Limbo R, Schroeder M. (Eds.). (2018). Guided participation in pediatric nursing practice: Relationship-based teaching and learning with parents, children, and adolescents. New York: Springer.